CLINICAL TRIAL: NCT05060744
Title: Study Off Efficacy and Rapidity of Action of a Product With Sodium Alginate, Calcium and Magnesium Salts, Hyaluronic Acid and Aloe Vera to Control Oesophageal-Gastric Acidity (pH), Symptoms of Gastric Reflux and Hyperacidity
Brief Title: Efficacy and Speed of Action of a Product to Control Gastric Hydration and Gastroesophageal Reflux
Acronym: AQUAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Uriach Consumer Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URI-AQUAA-2020-01
Record Dates: First submitted 2021-09-17; First posted 2021-09-29 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2022-10

CONDITIONS: Oesophageal Reflux; Gastric Reflux; Hyperactivity; Stomach
Keywords: Oesophageal Reflux; Gastric Reflux; Hyperactivity; Stomach; Sodium Alginate; Calcium; Magnesium Salts; Hyaluronic Acid; Aloe Vera; Gastroenterology
MeSH Terms: conditions — Gastroesophageal Reflux; Spasm

STUDY DESIGN:
Intervention Model Description: Clinical trial with CE marked medical device under normal conditions of use.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Antacid) (Active Comparator): An Antacid, a CE marked medical device under normal conditions of use.
  Sodium alginate (reduces reflux) (250 mg/tablet) Calcium carbonate (reduces acidity) (80 mg/tablet) Magnesium carbonate (reduces acidity) (144 mg/tablet) Hyaluronic acid (mucosal protector) (6.15 mg/tablet) Aloe vera extract without anthraquinones (mucosal protector) (40 mg/tablet)
  Patients should take 2 tablets of treatment at the time they develop reflux or hyperacidity. The maximum dose will be 6 tablets per day.
  Interventions: Device: Antacid
- Control (Placebo Comparator): The control will consist of a placebo based on excipients without active ingredients that will be formulated so that the tablet has the same appearance as the test product, with three different colour layers.
  Patients should take 2 tablets of treatment at the time they develop reflux or hyperacidity. The maximum dose will be 6 tablets per day.
  Interventions: Other: Control

INTERVENTIONS:
Device: Antacid — The tablets should be kept in the mouth without chewing or swallowing, allowing them to dissolve completely.
  Other Names: Aquilea Antacid
  Arms: Intervention (Antacid)
Other: Control — The tablets should be kept in the mouth without chewing or swallowing, allowing them to dissolve completely.
  Arms: Control

SUMMARY:
A Randomised, Placebo-Controlled Clinical Trial off the Efficacy and Rapidity of Action of a Product Containing Sodium Alginate, Calcium and Magnesium Salts, Hyaluronic Acid and Aloe Vera to Control Oesophageal-Gastric pH and Reduce Symptoms of Gastric Reflux and Hyperacidity.

DETAILED DESCRIPTION:
The investigators will include patients with gastroesophageal reflux disease and heartburn (more than 3 weekly episodes of heartburn for at least 4 consecutive weeks) not related to medication intake and don't use proton pump blockers or H2-receptor antagonists.

This is a multicentre clinical trial with two-phase design:

Phase I: A double-blind, randomised, placebo-controlled clinical trial to assess the efficacy and rapidity of action of the medical device to reduce clinical symptoms of gastric reflux and hyperacidity under normal conditions of use. This phase I will be performed in primary care clinics.

Phase II: A non-comparative, non-controlled clinical trial to objectively assess, using continuous pH monitoring, the magnitude and rapidity to control gastric and oesophageal pH after taking the product. This phase II will be performed at the Department of Gastroenterology of Medic Center.

The study will begin with the baseline visit (day 0) in which the inclusion and exclusion criteria will be confirmed, the signing of informed consent will be obtained, GERD-Q Questionnaire will be done and treatment will be prescribed, followed by a home recording where patients will record data on episodes of acidity and heartburn occuring during the follow-up week. A face-to-face visit will be at 7 days after to recollect information about total number of daytime and nighttime episodes of acidity/heartburn since the previous visit and repeat the GERD-Q Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes over 18 years of age
* Patients with gastroesophageal reflux disease and heartburn (more than 3 weekly episodes of heartburn for at least 4 consecutive weeks) not related to medication intake
* Patients not on proton pump blockers or H2-receptor antagonists
* Patients able to understand the study implications and who sign the informed consent.

Exclusion Criteria:

* Pregnant or nursing women
* Patients who are currently using or have used other medications or antacid products for the treatment of reflux and hyperacidity symptoms within 7 days prior to enrolment in this study.
* Patients treated with antihypertensive drugs, calcium channel blockers or non-steroidal anti-inflammatory drugs (NSAIDs)
* Patients with hypercalcaemia, hypertension, renal failure or other conditions in which the use of the components of the investigational product is not recommended.
* Patients with serious diseases that, in the physician's opinion, could interfere with the results of the study or prevent their participation in it.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-09 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Intensity of acidity/heartburn | At the beginning and at the end of treatment, an average of 7±1 days in patients
  Change in intensity of acidity/heartburn before and after taking the treatment, assessed by the patient using a visual analogue scale (VAS from 0=none to 10=maximum imaginable)
Time from treatment intake to resolution or maximum decrease in acidity/heartburn | At the beginning and at the end of treatment, an average of 7±1 days in patients
  Change in time from treatment intake to resolution or maximum decrease in acidity/heartburn as assessed by the patient using a 3-point Likert scale (<1 minute, 1-5 minutes, >5 minutes)
Time elapsed between product intake and intragastric pH > 4 | Baseline visit
  Change in minutes of the time elapsed between product intake and intragastric pH > 4
Time with intragastric pH > 4 for 20 minutes before and after product intake | Baseline visit
  Total time in minutes of the time in intragastric pH > 4 for 20 minutes before and after product intake

SECONDARY OUTCOMES:
Demographic data | Baseline visit
  Sex, ethnicity and age data of patients
Time of tablet duration in the mouth before complete dissolution | At the beginning and at the end of treatment, an average of 7±1 days in patients
  Change in time of tablet duration in the mouth before complete dissolution, assessed using a 4-point Likert scale (< 1 minute, 1-3 minutes, 3-5 min, >5 minutes)
Number of daytime and nightime episodes of acidity/heartburn | An average of 7±1 days in patients
  Change in number of daytime and nightime episodes of acidity/heartburn (information recorded in the Patient Diary)
Intensity of reflux before and after treatment | At the beginning and at the end of treatment, an average of 7±1 days in patients
  Change in intensity of reflux before and after treatment, assessed by the patient using a visual analogue scale (VAS from 0=none to 10=maximum imaginable)
Gastroesophageal Reflux Disease Questionnaire (GERD-Q) score | At the beginning and at the end of treatment, an average of 7±1 days in patients
  Change in Gastroesophageal Reflux Disease Questionnaire (GERD-Q) score. Between 0 and 8 in symptoms questions the score don't mean GERD, more than 8 mean GERD or severe GERD if in impact questions the score is more than 2.
Number of Participants With Adverse Events | From the beginning to the end of treatment, an average of 7±1 days in patients
  Number of Participants With Adverse Events as a Measure of Safety and Tolerability
Degree of physician and patient satisfaction with the efficacy, rapidity of action and tolerability of the product | Through study completion, an average of 6 months
  Assessment of degree of physician and patient satisfaction with the efficacy, rapidity of action and tolerability of the product using 5-point Likert scales (0=very dissatisfied, 1=dissatisfied, 2=indifferent, 3=satisfied, 4=very satisfied).
Mean intragastric pH | Baseline visit
  Change in mean intragastric pH for 20 minutes before and after product intake
Number of episodes of GER (intraoesophageal pH < 4) | Baseline visit
  Change in the number of episodes of GER (intraoesophageal pH < 4). Evaluation 20 minutes before and after taking the product
Time with oesophageal pH < 4 | Baseline visit
  Change in the time with oesophageal pH < 4. Evaluation 20 minutes before and after taking the product
Longest reflux episode (oesophageal pH <4) | Baseline visit
  Change in the time of longest reflux episode (oesophageal pH <4). Evaluation 20 minutes before and after taking the product

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Armengol, Ph, Principal Investigator — Primary Health Center Poblenou, Barcelona, Spain
Locations (1):
- Oriol Armengol, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No